CLINICAL TRIAL: NCT02784418
Title: SHam-controlled INtErvention to Improve QOL in CTOs: the SHINE CTO Trial
Brief Title: The SHINE-CTO Trial
Acronym: SHINE-CTO
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues due to the pandemic
Sponsor: Minneapolis Heart Institute Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16-009
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion of Coronary Artery; Percutaneous Transluminal Coronary Angioplasty
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI of CTO (Active Comparator): Intervention: PCI of CTO (Chronic Total Occlusion Percutaneous Coronary Intervention) Chronic Total Occlusion Percutaneous Coronary Intervention (CTO PCI), as per standard clinical practice. Hospitalized overnight after the procedure, with post procedure monitoring practices as per standard of care for PCI. CTO PCI patients will receive blinded clopidogrel 75 mg daily for 6 months.
  Interventions: Procedure: Chronic Total Occlusion Percutaneous Coronary Intervention
- Sham Procedure (Sham Comparator): Intervention: Sham procedure Subjects will be blinded to randomization assignment using a combination of conscious sedation and sensory isolation (e.g., blindfold and noise isolation). Control subjects will only undergo a "Sham procedure", wherein they will undergo bilateral arterial access, without angiography or PCI being performed. Hospitalized overnight after the procedure, with post procedure monitoring practices as per standard of care for PCI. Sham group will receive blinded placebo clopidogrel for 6 months.
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Procedure: Chronic Total Occlusion Percutaneous Coronary Intervention — Chronic Total Occlusion Percutaneous Coronary Intervention (CTO PCI), as per standard clinical practice
  Arms: PCI of CTO
Procedure: Sham Procedure — Sham Procedure: Bilateral arterial access, without angiography or PCI being performed
  Arms: Sham Procedure

SUMMARY:
Design: Single center, double-blind, sham-controlled trial that will randomize symptomatic patients with a coronary chronic total occlusion (CTO) to CTO percutaneous coronary intervention (PCI) or a sham procedure. All patients will receive optimal medical therapy.

Treatment:CTO PCI, as per standard clinical practice.

Control: Patients randomized to sham-procedure will undergo only bilateral arterial access, without angiography or PCI being performed.

Secondary Endpoints: (1) Greater improvement in SAQ-7 Summary scores during the entire duration of follow-up (6 months) using a repeated measures analysis (2) Greater improvement in individual components of patients' health status (3) Greater improvement in exercise capacity (4) Similar incidence of major adverse cardiac events (MACE), both peri-procedural and long-term

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Willing and able to give informed consent. The patients must be able to comply with study procedures and follow-up.
* Referred for clinically-indicated CTO PCI
* Optimal medical therapy (at least two anti-anginal medications at maximum tolerated doses, aspirin, and statin)

Exclusion Criteria:

* Coexisting conditions that limit life expectancy to less than 6 months or that could affect a patient's compliance with the protocol
* Recent (<7 days) acute myocardial infarction
* Patient has no symptoms related to the CTO
* Known allergy to aspirin or clopidogrel
* Increased risk of bleeding (need for warfarin, oral Xa inhibitor, or thrombin inhibitor administration, recent [within 30 days] major bleed, known bleeding diathesis or coagulation disorder)
* Positive pregnancy test or breast-feeding
* Chronic kidney disease, defined as serum creatinine > 2.5 mg/dL
* Severe peripheral arterial disease limiting exercise capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Greater improvement in disease-specific health status, as assessed by the 7-item Seattle Angina Questionnaire (SAQ) Summary Score (SAQ-7, an established measure of health status in patients with coronary artery disease) | 1 month

SECONDARY OUTCOMES:
Greater improvement in SAQ-7 Summary scores during the entire duration of follow-up using a repeated measures analysis | 6 months
Greater improvement in individual components of patients' health status, as assessed by the SAQ Physical Limitation, Angina Frequency, and Quality of Life domains of the SAQ-7 score | Baseline and 6 months
Greater improvement in individual components of patients' health status, as assessed by the EuroQol-5D (EQ-5D) | Baseline and 6 months
Greater improvement in individual components of patients' health status, as assessed by the Rose Dyspnea Score | Baseline and 6 months
Greater improvement in exercise capacity, as assessed by treadmill exercise stress | Prior to and 1 month after index procedure
Similar incidence of major adverse cardiac events (MACE), both peri-procedural and long-term | 6 months
Favorable incremental cost-effectiveness ratio | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Study Chair — Minneapolis Heart Institute

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brilakis ES, Grantham JA, Rinfret S, Wyman RM, Burke MN, Karmpaliotis D, Lembo N, Pershad A, Kandzari DE, Buller CE, DeMartini T, Lombardi WL, Thompson CA. A percutaneous treatment algorithm for crossing coronary chronic total occlusions. JACC Cardiovasc Interv. 2012 Apr;5(4):367-79. doi: 10.1016/j.jcin.2012.02.006. PMID 22516392
- [Background] Kahn JK. Angiographic suitability for catheter revascularization of total coronary occlusions in patients from a community hospital setting. Am Heart J. 1993 Sep;126(3 Pt 1):561-4. doi: 10.1016/0002-8703(93)90404-w. PMID 8362709
- [Background] Christofferson RD, Lehmann KG, Martin GV, Every N, Caldwell JH, Kapadia SR. Effect of chronic total coronary occlusion on treatment strategy. Am J Cardiol. 2005 May 1;95(9):1088-91. doi: 10.1016/j.amjcard.2004.12.065. PMID 15842978
- [Background] Werner GS, Gitt AK, Zeymer U, Juenger C, Towae F, Wienbergen H, Senges J. Chronic total coronary occlusions in patients with stable angina pectoris: impact on therapy and outcome in present day clinical practice. Clin Res Cardiol. 2009 Jul;98(7):435-41. doi: 10.1007/s00392-009-0013-5. Epub 2009 Mar 18. PMID 19294443
- [Background] Grantham JA, Jones PG, Cannon L, Spertus JA. Quantifying the early health status benefits of successful chronic total occlusion recanalization: Results from the FlowCardia's Approach to Chronic Total Occlusion Recanalization (FACTOR) Trial. Circ Cardiovasc Qual Outcomes. 2010 May;3(3):284-90. doi: 10.1161/CIRCOUTCOMES.108.825760. Epub 2010 Apr 13. PMID 20388873
- [Background] Joyal D, Afilalo J, Rinfret S. Effectiveness of recanalization of chronic total occlusions: a systematic review and meta-analysis. Am Heart J. 2010 Jul;160(1):179-87. doi: 10.1016/j.ahj.2010.04.015. PMID 20598990